CLINICAL TRIAL: NCT04292015
Title: Impact of Retinopathy of Prematurity Screening Examination on Cardiorespiratory Indices - A Comparison of Optos Ultra-Widefield Retinal Imaging and Binocular Indirect Ophthalmoscopy
Brief Title: Optos Versus Indirect Ophthalmoscopy for ROP Screening Examination (Optos vs BIO Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: DHRD/2017/043
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Pre-Term
Keywords: opthalmology; neonatal; premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Each premature infant recruited into the study will undergo retinal imaging with the Optos ultra-widefield retinal imaging device as well as the gold standard method of examination with the binocular indirect ophthalmoscope. The order of the procedures to be carried out in each infant will be determined by randomisation via sealed envelopes prepared remotely by a member of the pilot team not involved in the recruitment of patients or their screenings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard then Intervention (Experimental): Infant will undergo standard method of examination with binocular indirect opthalmoscope (BIO) followed by retinal imaging with Optos ultra-wide field retinal imaging device.
  Interventions: Diagnostic Test: Optos ultra-widefield retinal imaging (Optos California)
- Intervention then Standard (Experimental): Infant will undergo retinal imaging with Optos ultra-wide field retinal imaging device followed by standard method of examination with binocular indirect opthalmoscope (BIO).
  Interventions: Diagnostic Test: Optos ultra-widefield retinal imaging (Optos California)

INTERVENTIONS:
Diagnostic Test: Optos ultra-widefield retinal imaging (Optos California) — retinal imaging device

SUMMARY:
ROP is a preventable cause of blindness in premature infants. It is routinely screened for by using an indirect ophthalmoscope, a scleral depressor, and a condensing lens. This method of screening can cause significant cardiorespiratory distress to infants. A new camera (Optos California) has recently been used to image infants with different severities of ROP. The Optos California is capable of capturing up to 200 degrees of retina in a single image without contact with the eye. The non eye contact nature of the Optos California may cause less distress to infants who are due a ROP screening examination. The present study is to compare the impact of ROP screening examination between the Optos retinal camera and conventional binocular indirect ophthalmoscopy using cardiorespiratory indices (such as heart rate, oxygen saturations, blood pressure, and respiratory rate) as a measure of distress.

DETAILED DESCRIPTION:
This is a pilot prospective randomised study. As part of the routine clinical care at RDH, all premature infants eligible for ROP screening as stated by the UK ROP screening guidelines will undergo the gold standard screening examination by a Consultant Ophthalmologist.

Each infant eligible for ROP screening will be routinely scheduled for several ROP screening examinations prior to discharge from the neonatal unit. For each infant who is eligible and whose parent(s) or legal guardian have agreed for them to be enrolled in the study, two additional procedures to the gold standard examination with the binocular indirect ophthalmoscope (as stated above) will be carried out at each of its routinely scheduled ROP screening examination.

The first additional procedure will be the acquisition of images of both fundi by Ophthalmology Specialty Registrar with the Optos ultra-widefield retinal-imaging device. Cardiorespiratory indices will be collected at different time points of the Optos retinal imaging procedure.

The second additional procedure will be the collection of cardiorespiratory indices (including the heart rate,respiratory rate, oxygen saturations, and blood pressure) by the paediatric research nurse at the time of the gold standard examination with the binocular indirect ophthalmoscope. The equipment used will be the same as those used to measure the cardiorespiratory indices during different time points of the Optos ultra-widefield retinal imaging procedure (see above).

ELIGIBILITY:
Inclusion Criteria:

* Infants eligible for routine ROP screening using UK ROP screening guidelines (Any infant born at or before 32 weeks gestation and/or weigh 1500 grams or less).
* Infants with parents who have conversational English and who can give written informed consent.

Exclusion Criteria:

* Infants not eligible for routine ROP screening under UK ROP screening guidelines.
* Infants who are deemed not well enough by a consultant neonatologist (SO) for retinal examination or retinal imaging.
* Any premature infant with media opacities that prevents adequate visualisation of the retina.
* Inability of the parents to understand verbal and written English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Blood pressure (BP) | Baseline to 10 minutes following completion of both interventions
  Blood pressure (BP)
Number of infants that develop bradycardia | Baseline to 10 minutes following completion of both interventions
  Defined as less than 100 beats per minute
Oxygen saturation | Baseline to 10 minutes following completion of both interventions
  Number of infants who develop oxygen saturations below 85%
Development of respiratory distress | Baseline to 10 minutes following completion of both interventions
  Number of infacnts who develop respiratory distress, defined as respiratory rate less than 30 breaths per minute

SECONDARY OUTCOMES:
Determine and compare time taken to perform interventions | During intervention
  Time of each intervention recorded

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Derby & Burton NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No